CLINICAL TRIAL: NCT02816645
Title: One-year Follow-up of Iron in Basal Ganglia - R2*: a Biomarker of Parkinson's Disease Progression?
Acronym: MPI-R2*
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: France Parkinson Association (Other); Federation for Brain Research (Unknown); NS-PARK Network (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0268; 2014-A01184-43 (Other: 2014-A01184-43)
Record Dates: First submitted 2016-06-20; First posted 2016-06-28 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Biomarker; Iron; R2*; MRI; Patients; UK Parkinson's Disease Society Brain Bank
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Spectroscopy

ARMS (4):
- <5 years (Experimental): 160 PD patients divided into four subgroups of 40 patients according to disease duration:
  * < 5 years
  * Between 5 and 10 years
  * Between 10 and 15 years
  * > 15 years
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)
- Between 5 and 10 years (Experimental): 160 PD patients divided into four subgroups of 40 patients according to disease duration:
  * < 5 years
  * Between 5 and 10 years
  * Between 10 and 15 years
  * > 15 years
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)
- Between 10 and 15 years (Experimental): 160 PD patients divided into four subgroups of 40 patients according to disease duration:
  * < 5 years
  * Between 5 and 10 years
  * Between 10 and 15 years
  * > 15 years
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)
- > 15 years (Experimental): 160 PD patients divided into four subgroups of 40 patients according to disease duration:
  * < 5 years
  * Between 5 and 10 years
  * Between 10 and 15 years
  * > 15 years
  Interventions: Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI)

SUMMARY:
The study of non-invasive and reliable biomarkers to track progression of Parkinson's disease (PD) is essential while disease-modifying treatments are being developed. Many clinical biological or imaging biomarkers have been tested but no "gold standard" has been found as of yet. Among these, Magnetic Resonance Imaging (MRI) relaxometry using R2* measurement (R2* = 1/T2*), which is a validated marker for estimating brain iron concentration, appears to be an attractive technique because its safety, rapidly measured in clinical conditions and its ease to ensure individual longitudinal follow-up. Current data of cross sectional studies of R2*, which have shown an iron increase in Substantia Nigra (SN), led to suppose that it could be a biomarker of disease vulnerability. Recently, the investigators have conducted the first longitudinal follow-up of R2* (1.5 T MRI), which showed a rapid R2* increase in both parts of the SN and in the caudal putamen. We propose, here, a multicenter prospective study of one-year cohort follow-up of R2* variations (ΔR2*) in three regions of interest (ROIs) (the SN, the Ventral Tegmental Area (VTA) and the Putamen) of 160 patients with PD, using a 3 Tesla MRI, to evaluate the potential interest of R2* as a biomarker of disease progression. The variation of R2* (ΔR2*) will be correlated with clinical markers of disease progress, non-motor symptoms. 80 healthy controls subjects will also be included to assess the effect of aging on cerebral physiological iron levels.

DETAILED DESCRIPTION:
Use lay language.

The study of non-invasive and reliable biomarkers to track progression of Parkinson's disease is essential while disease-modifying treatments are being developed. Many clinical biological or imaging biomarkers have been tested but no "gold standard" has been found as of yet. Among these, Magnetic Resonance Imaging (MRI) relaxometry using R2* measurement (R2* = 1/T2*), which is a validated marker for estimating brain iron concentration, appears to be an attractive technique because its safety, rapidly measured in clinical conditions and its ease to ensure individual longitudinal follow-up. Current data of cross sectional studies of R2*, which have shown an iron increase in substantia nigra, led to suppose that it could be a biomarker of disease vulnerability. Recently, we have conducted the first longitudinal follow-up of R2* (1.5 T MRI), which showed a rapid R2* increase in both parts of the SN and in the caudal putamen. We propose, here, a multicenter prospective study of one-year cohort follow-up of R2* variations (ΔR2*) in three regions of interest (the substantia nigra, the ventral tegmental area and the putamen) of 160 patients with Parkinson's disease, using a 3 Tesla MRI, to evaluate the potential interest of R2* as a biomarker of disease progression. The variation of R2* (ΔR2*) will be correlated with clinical markers of disease progress, non-motor symptoms. 80 healthy controls subjects will also be included to assess the effect of aging on cerebral physiological iron levels.

Type of study : Interventional multicenter prospective study of cohort follow-up.

Number of centers : 6 (Clermont-Ferrand, Lyon, Grenoble, Paris, Limoges, Lille)

Study population :

Recruitment

160 patients with Parkinson's disease divided into four subgroups of 40 patients according to disease duration:

* < 5 years
* Between 5 and 10 years
* Between 10 and 15 years
* > 15 years

In parallel, 80 sex-age matched healthy controls subjects matched equally distributed in the 4 groups (n = 20/group) based on a stratified plan by gender and age (ratio 1:2).

Subjects will be assessed twice, one year apart by the procedures detailed below. The two neurological assessments should be made by the same certified neurologist.

Patients' procedure:

Visit 1 (Day 0) (duration: 1 day or 2 half days)

* Signature of an informed consent form (only at Day 0).
* Demographic and clinical characteristics (sex, age, disease duration, treatments).
* Neurological evaluation.
* Neuropsychological evaluation.
* Self-administered questionnaires.
* 1st MRI acquisition.

Visit 2 (Day 0 + 1 year) (duration: 1 day or 2 half days)

* Current treatment(s), adverse event(s), serious adverse event(s).
* Neurological evaluation.
* Neuropsychological evaluation.
* Self-administered questionnaires.
* 2d MRI acquisition.

Matched healthy controls subjects' procedure:

Visit 1 (Day 0) (duration: 1 half day)

* Signature of an informed consent form (only at Day 0).
* Demographic and clinical characteristics (sex, age, disease duration, treatments).
* Brief neuropsychological evaluation.
* 1st MRI acquisition.

Visit 2 (Day 0 + 1 year) (duration: 1 half day)

* Current treatment(s), adverse event(s), serious adverse event(s).
* Brief neuropsychological evaluation.
* 2d MRI acquisition.

MRI acquisition (duration: 45 to 60 min)

The procedure will be performed on a 3 Tesla MRI, allowing a substantial gain in signal-to-noise ratio compared with the one obtained at 1.5 Tesla.

Different sequences will be planned:

* T2-weighted sequence * 3D GRE multi-echo. This sequence will generate a R2* maps of the whole brain.
* T1-weighted sequence in high resolution 3D. This sequence will allow the anatomical characterization of different brain structures and will help the normalization of T2* in pictures an anatomical reference space.
* T2* sequence 3D multiple gradient echo (Spoiled Gradient Recalled echo sequence). This sequence will measure the decay rate of NMR signal according to the echo time.
* 2D spin echo sequence T1-weighted for neuromelanin. This sequence view the substantia nigra and locus coeruleus (optional sequence).
* Optional Diffusion-weighted sequence. This sequence determines the movements of water molecule in the brain and to infer the main lines of connections between neurons (optional sequence).

The R2* (1/T2*) will be measured in three different regions of interest (substantia nigra, ventral tegmental area and the putamen) for the 2 MRI's in order to calculate ΔR2.

ELIGIBILITY:
Inclusion criteria for PATIENTS :

* Parkinson's Disease (UK Parkinson's Disease Society Brain Bank Criteria).
* No Deep Brain Stimulation (DBS).
* From 40 to 80 years old.

Inclusion criteria for HEALTHY CONTROL SUBJECTS :

- From 40 to 80 years old.

Exclusion criteria for PATIENTS :

* Dementia (MoCA < 24).
* Atypical parkinsonism (MSA, PSP, …).
* Severe current psychiatric or somatic disease.
* Iron treatments (Desferal® (deferoxamine), Ferriprox® (deferiprone) et Exjade® (deferasirox), Fumafer® (ferrous fumarate), Tardyferon® (ferrous sulfate (II)),…), Ferinject® (ferric carboxymaltose), Venofer® (iron sucrose),…).
* Contra-indication to MRI (claustrophobia, pace maker,…).

Exclusion criteria for HEALTHY CONTROL SUBJECTS :

* Neurological disease.
* Psychiatric or somatic disease.
* Dementia (MoCA < 24).
* Iron treatments (Desferal® (deferoxamine), Ferriprox® (deferiprone) et Exjade® (deferasirox), Fumafer® (ferrous fumarate), Tardyferon® (ferrous sulfate (II)),…), Ferinject® (ferric carboxymaltose), Venofer® (iron sucrose),…).
* Contra-indication to MRI (claustrophobia, pace maker,…).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline cerebral R2* | at 1 year
  Change from baseline cerebral R2* quantification at 1 year in three regions of interest (Substantia Nigra, Ventral Tegmental Area and Putamen).

SECONDARY OUTCOMES:
Change from baseline Parkinson's disease clinical symptoms | at 1 year
  - Change from baseline Parkinson's disease clinical symptoms at one year with the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS Score.
Change from baseline severity of Parkinson's disease | at 1 year
  - Change from baseline severity of Parkinson's disease at one year with the HOEHN & YAHR status.
Change from baseline activities of daily living | at 1 year
  - Change from baseline activities of daily living at one year with the SCHWAB & ENGLAND scale.
Change from baseline freezing | at 1 year
  - Change from baseline freezing at one year with the Freezing of Gait Questionnaire (FOG-Q).
change from baseline cognitive function | at 1 year
  - Change from baseline cognitive function at one year with the Montreal Cognitive Assessment (MoCA).
Change from baseline hyper and hypo dopaminergic symptoms scores | at 1 year
  - Change from baseline hyper and hypo dopaminergic symptoms scores at one year with the Ardouin Scale of Behavior in Parkinson's Disease (ASBPD)
Change from baseline sleepiness score | at 1 year
  Change from baseline sleepiness score at one year with the Epworth Sleepiness Scale (ESS).
Change from baseline autonomic functions score | at 1 year
  Change from baseline autonomic functions score at one year with the SCales for Outcomes in Parkinson's disease (SCOPA-AUT).
Change from baseline non-motor symptoms score | at 1 year
  Change from baseline non-motor symptoms score at one year with the Non-Motor symptom assessment Scale for Parkinson's Disease (NMSS).
Change from baseline apathy score | at 1 year
  - Change from baseline apathy score at one year with the Lille Apathy Rating Scale (LARS).
Change from baseline depression score | at 1 year
  - Change from baseline depression score at one year with the Hamilton Rating Scale for Depression (HAM-D).
Change from baseline anxiety score | at 1 year
  - Change from baseline anxiety score at one year with the Hamilton Rating Scale for Anxiety (HAM-A).

CONTACTS AND LOCATIONS:
Overall Officials: Anna MARQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (13):
- France (13):
  - Chu Pellegrin, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - Chu Lille, Lille
  - Chu Dupuytren, Limoges
  - Hôpital neurologique Pierre Wertheimer, Lyon
  - Chu Montpellier, Montpellier
  - Chu Nancy, Nancy
  - CHU Pitié Salpétrière, Paris
  - Hôpital Henri Mondor, Paris
  - Chu Poitiers, Potiers
  - Chu Reims, Reims
  - Chu Toulouse, Toulouse